CLINICAL TRIAL: NCT03421379
Title: A Phase 3 Study of Nasal Glucagon (LY900018) Compared to Intramuscular Glucagon for Treatment of Insulin-induced Hypoglycemia in Japanese Patients With Diabetes Mellitus
Brief Title: A Study of Nasal Glucagon (LY900018) in Japanese Participants With Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16962; I8R-JE-IGBJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Glucagon Nasal Powder (Experimental): A single dose of 3 milligram (mg) glucagon nasal powder administered intranasally.
  Interventions: Drug: Glucagon Nasal Powder
- Glucagon Hydrochloride Solution (Active Comparator): A single dose of 1 mg glucagon hydrochloride solution was administered intramuscular (IM)
  Interventions: Drug: Glucagon Hydrochloride Solution

INTERVENTIONS:
Drug: Glucagon Nasal Powder — Administered intranasally
  Other Names: LY900018
  Arms: Glucagon Nasal Powder
Drug: Glucagon Hydrochloride Solution — Administered IM
  Other Names: GlucaGen®
  Arms: Glucagon Hydrochloride Solution

SUMMARY:
The purpose of this study is to determine the efficacy and safety of nasal glucagon compared to intramuscular (IM) glucagon for treatment of insulin-induced hypoglycemia in Japanese participants with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Type 1 diabetes (T1D) or Type 2 diabetes (T2D)
* Body mass Index (BMI) of 18.5 to 30.0 kilograms per meter squared (kg/m2) for T1D, or 18.5 to 35.0 kg/m2 for T2D
* Hemoglobin A1c (HbA1c) ≤10%

Exclusion Criteria:

* Have significant changes in insulin regimen and/ or unstable blood sugar control within the past 3 month
* Have received a total daily dose of insulin >1.2 units per kilogram (U/kg)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Japan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Seaquist E, Gimenez M, Yan Y, Matsuhisa M, Kao CY, Wadwa RP, Nagai Y, Khunti K. Nasal Glucagon Reverses Insulin-induced Hypoglycemia With Less Rebound Hyperglycemia: Pooled Analysis of Clinical Trials. J Endocr Soc. 2024 Feb 26;8(4):bvae034. doi: 10.1210/jendso/bvae034. eCollection 2024 Feb 19. PMID 38444629

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive either nasal glucagon or intramuscular (IM) glucagon in the first period, followed by the alternate treatment in the second period.
Groups:
- Glucagon Nasal Powder/Glucagon Hydrochloride: A single dose of 3 milligram (mg) glucagon nasal powder was administered intranasally in period 1 then 1 mg single dose intramuscular glucagon hydrochloride solution was administered in period 2.
- Glucagon Hydrochloride Solution/Glucagon Nasal Powder: A single dose of 1 mg glucagon hydrochloride solution was administered intramuscular (IM) in period 1 then 3 mg single dose glucagon nasal powder was administered in period 2.
Period: Period 1
Arm/Group | Glucagon Nasal Powder/Glucagon Hydrochloride | Glucagon Hydrochloride Solution/Glucagon Nasal Powder
Started | 34 | 41
Received at Least One Dose of Study Drug | 33 | 39
Completed | 32 | 37
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Did not receive treatment | 1 | 2
Period: Washout Period (3 to 14 Days)
Arm/Group | Glucagon Nasal Powder/Glucagon Hydrochloride | Glucagon Hydrochloride Solution/Glucagon Nasal Powder
Started | 32 | 37
Completed | 32 | 37
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Glucagon Nasal Powder/Glucagon Hydrochloride | Glucagon Hydrochloride Solution/Glucagon Nasal Powder
Started | 32 | 37
Completed | 32 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Glucagon Nasal Powder/Glucagon Hydrochloride Solution: A single dose of 3 mg glucagon nasal powder was administered intranasally
- Glucagon Hydrochloride Solution/Glucagon Nasal Powder: A single dose of 1 mg glucagon hydrochloride solution was administered IM
- Total: Total of all reporting groups
Arm/Group | Glucagon Nasal Powder/Glucagon Hydrochloride Solution | Glucagon Hydrochloride Solution/Glucagon Nasal Powder | Total
Number analyzed (Participants) | 33 | 39 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.6) | 57.5 (9.2) | 50.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 20 | 30 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 39 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 33 | 39 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 33 | 39 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Treatment Success During Controlled Insulin-Induced Hypoglycemia
Description: Percentage of participants who achieved treatment success during the controlled insulin-induced hypoglycemia in participants with type 1 diabetes mellitus (T1DM) and participants with type 2 diabetes mellitus (T2DM).Treatment success is defined as an increase in plasma glucose to greater than or equal to (≥) 70 milligrams per deciliter (mg/dL) or an increase of ≥20 mg/dL from plasma glucose nadir, without receiving additional actions to increase the plasma glucose concentration. Nadir is defined as the minimum plasma glucose concentration at the time of or within 10 minutes following glucagon administration.
Time Frame: Pre-dose up to 30 minutes post each glucagon administration
Population: All randomized participant who completed both treatment visits and had evaluable treatment success data.
Measure: Number; unit: percentage of participants
Groups:
- Glucagon Nasal Powder: A single dose of 3 mg glucagon nasal powder was administered intranasally
- Glucagon Hydrochloride Solution: A single dose of 1 mg glucagon hydrochloride solution was administered IM
Arm/Group | Glucagon Nasal Powder | Glucagon Hydrochloride Solution
Number analyzed (Participants) | 68 | 68
percentage of participants | 100 | 100
Statistical Analysis 1: Comparison: Glucagon Nasal Powder vs Glucagon Hydrochloride Solution; Test type: Non-Inferiority — The pre-defined non-inferiority margin is (10%); Treatment Difference Wald's Method = 0.00, 95% CI 2-sided [-1.47 to 1.47]

2. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Maximal Blood Glucose (BGmax) of Glucagon Nasal Powder and Glucagon Hydrochloride Intramuscular (IM)
Description: PD assessment measured the change from Baseline in maximal blood glucose (BGmax) of Glucagon Nasal Powder and Glucagon Hydrochloride intramuscular (IM).
Time Frame: Pre-dose, 5, 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, 240 minutes after each glucagon administration
Population: All randomized patients who receive at least 1 dose of the study drug and have evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram/deciliter (mg/dL)
Arm/Group | Glucagon Nasal Powder | Glucagon Hydrochloride Solution
Number analyzed (Participants) | 71 | 70
milligram/deciliter (mg/dL) | 113 (32) | 119 (33)

3. Secondary Outcome: PD: Time to Maximal Concentration (Tmax) of Glucagon Nasal Powder and Glucagon Hydrochloride IM
Description: PD assessment measured the time to maximal concentration (Tmax) of Glucagon Nasal Powder and Glucagon Hydrochloride IM.
Time Frame: Pre-dose, 5, 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, 240 minutes after each glucagon administration
Population: All randomized participants who received at least one dose of study drug and had evaluable PD data.
Measure: Median (Full Range); unit: hour
Arm/Group | Glucagon Nasal Powder | Glucagon Hydrochloride Solution
Number analyzed (Participants) | 71 | 70
hour | 1.00 [0.50 to 4.02] | 1.50 [0.67 to 4.00]

4. Secondary Outcome: Pharmacokinetics (PK): Change From Baseline in Area Under the Concentration Versus Time Curve From Zero to Time t (AUC [0-tLast]) of Glucagon Nasal Powder and Glucagon Hydrochloride IM
Description: PK assessment measured the change from baseline in the area under the concentration versus time curve from time zero to time t, where t is the last time point with a measurable concentration of Glucagon Nasal Powder and Glucagon Hydrochloride IM.
Time Frame: Pre-dose, 5, 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, 240 minutes after each glucagon administration
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hour/milliliter (pg*h/mL)
Arm/Group | Glucagon Nasal Powder | Glucagon Hydrochloride Solution
Number analyzed (Participants) | 71 | 68
Picogram*hour/milliliter (pg*h/mL) | 4830 (89) | 3240 (32)

5. Secondary Outcome: PK: Change From Baseline in Maximal Concentration (Cmax) of Glucagon Nasal Powder and Glucagon Hydrochloride IM
Description: PK assessment measured the change from baseline in maximal concentration (Cmax) of glucagon nasal powder and glucagon hydrochloride IM.
Time Frame: Pre-dose, 5, 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, 240 minutes after each glucagon administration
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/milliliter (pg/mL)
Arm/Group | Glucagon Nasal Powder | Glucagon Hydrochloride Solution
Number analyzed (Participants) | 71 | 68
picogram/milliliter (pg/mL) | 9520 (103) | 3290 (37)

6. Secondary Outcome: PK: Change From Baseline in Tmax of Glucagon Nasal Powder and Glucagon Hydrochloride IM
Description: PK assessment measured the change from baseline in Tmax of Glucagon Nasal Powder and Glucagon Hydrochloride IM.
Time Frame: Pre-dose, 5, 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, 240 minutes after each glucagon administration
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Glucagon Nasal Powder | Glucagon Hydrochloride Solution
Number analyzed (Participants) | 71 | 68
hour (h) | 0.25 [0.17 to 0.67] | 0.17 [0.08 to 0.67]

ADVERSE EVENTS:
Time Frame: From Baseline to End of Follow-up (Up to 2 Months)
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Glucagon Nasal Powder | Glucagon Hydrochloride Solution
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/71 | 1/70
Other Adverse Events (participants affected / at risk) | 15/71 | 13/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucagon Nasal Powder (N=71) | Glucagon Hydrochloride Solution (N=70)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucagon Nasal Powder (N=71) | Glucagon Hydrochloride Solution (N=70)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 11 (11)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03421379/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT03421379/SAP_001.pdf